CLINICAL TRIAL: NCT00826852
Title: Phase II Trial of Weekly Docetaxel and Four Weekly Carboplatin Combination in the First-line Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: Weekly Docetaxel and Four Weekly Carboplatin in Non-small Cell Lung Cancer Carbo-Tax
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976B_6020
Record Dates: First submitted 2008-10-13; First posted 2009-01-22 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel and carboplatin — weekly docetaxel 30mg/m2 and four weekly carboplatin AUC (Area under curve) 5

SUMMARY:
The purpose of this study is:

* to assess the efficacy of the combination in terms of Objective (clinical and radiological) Response Rate
* to assess the time to progression of the disease; assess the safety profile of the combination, and assess the survival time.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed inoperable locally advanced or metastatic non-small cell lung cancer
* ECOG Performance Status is 0-2
* At least one measurable lesion in two dimensions by means of CT scan
* No brain metastases
* No prior chemotherapy for this malignancy,
* Acceptable hematological profile (as defined by a leukocyte count ≥ 3000/mm3, a platelet count ≥ 100.000mm3 and Hb ≥ 9g/100mL), and adequate renal function (as defined by serum creatinine ≤ 1.5mg/dl or creatinine clearance measured in 24 hours urine ≥ 60 mL/min), and hepatic function (as defined by bilirubin ≤ 1.5 x maximum normal value even with hepatic metastasis; transaminases (ALT, AST) ≤ 2.5 x maximum normal value; alkaline phosphatase ≤ 2.5 x maximum normal value, except in case of a bone metastasis)

Exclusion Criteria:

* Concomitant use of another anti-cancer therapy
* Chemotherapy, radiotherapy or curative surgery
* Evidence of intracerebral metastasis
* Unstable medical condition that makes the patient to take part in a clinical study (congestive heart failure, serious arrhythmia, uncontrolled diabetes mellitus), history of myocardial infarction within last 3 months, massive pleural or peritoneal effusion; or presence of serious uncontrolled infection, diarrhea, ileus, interstitial pneumonia, pulmonary fibrosis.
* Presence of other tumours different from basal cell carcinoma of the skin, with disease free survival less then 3 years.
* Pregnancy or breastfeeding. In women of childbearing potential and in men, an adequate contraceptive method must be used
* Social or psychological condition that render the patient inadequate for the follow-up of the study
* Contraindication for any of the study drugs (e.g. history of hypersensitivity to any of the ingredients of the study drugs)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2003-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Efficacy by response rate | After the 3rd cycle, 6th cycle and at every follow up visit

SECONDARY OUTCOMES:
Adverse events | At each visit
Efficacy by time to progression | Until the progression of all patients
Overall survival | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)